CLINICAL TRIAL: NCT03494946
Title: A Randomized Clinical Trial Comparing Overall Survival in Selected Patients With ColoRectal Carcinoma Treated by Liver Transplantation or Chemotherapy
Brief Title: Liver Transplantation Compared to Chemotherapy in Patients With ColoRectal Cancer
Acronym: SECAIII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Smedman, MD, Consultant, gastrointestinal oncology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1657 SECAIII
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Liver Metastases; Colorectal Cancer
Keywords: Liver metastasis; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liver Transplantation; Drug Therapy

STUDY DESIGN:
Intervention Model Description: A randomized study were half of the subjects will be given standard chemo therapy and the other half will undergo liver transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Patients that suffer from Colorectal cancer and metastasis to liver that are randomized to Group A, will undergo Liver transplantation
  Interventions: Procedure: Liver transplantation
- Arm B (Active Comparator): Patients that suffer from Colorectal cancer and metastasis to liver that are randomized to Group B, will be given chemotherapy, TACE, SIRT or other available treatment options.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Liver transplantation
  Arms: Arm A
Drug: Chemotherapy — May include chemotherapy, TACE, SIRT or other available treatment options.
  Other Names: Other treatment
  Arms: Arm B

SUMMARY:
The trial is a randomized control trial. Patients are randomized between Ltx and other treatment that may include further chemotherapy, TACE, SIRT or other available treatment options. The patients will be randomized 1:1 to Ltx and chemotherapy/other treatment options.

DETAILED DESCRIPTION:
Patients with non-resectable CRC liver metastases evaluated at the liver MDT at Oslo University Hospital, Rikshospitalet will be included in the study. Patients should have progressive disease on 1.line chemotherapy or the treatment should have been stopped due to toxicity. Patients randomized to Ltx will if applicable stop bevazicumab. All patients (both arms) will start further treatment that may include chemotherapy, TACE, SIRT or other available treatment options. Patients not receiving a donor liver graft within 3 months after listing for transplantation will be taken off the waiting list and transferred to the chemotherapy/other treatment option group. Patients randomized to Ltx and developing progressive disease beyond the inclusion/exclusion criteria during the time on the waiting list will be excluded from the study and receive best treatment option at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma in colon/rectum.
* Liver metastases, not amenable to liver resection
* No signs of extra hepatic metastatic disease or local recurrence according to PET/CT scan within 6 weeks prior to the faculty meeting at the transplant unit, except patients may have resectable lung lesions all < 15mm.
* No signs of extra hepatic metastatic disease on CT or MRI thorax/abdomen/pelvis within 6 weeks prior to the faculty meeting at the transplant unit, except resectable lung lesions all < 15mm.
* No signs of extra hepatic metastatic disease on PET/CT within 6 weeks prior to the faculty meeting at the transplant unit, except patients may have resectable lung lesions all < 15mm
* Good performance status, ECOG 0 or 1.
* Satisfactory blood tests Hb >10g/dl, neutrophiles >1.0 (after any G-CSF), TRC >75, Bilirubin<1.5 x upper normal level, ASAT, ALAT<5 x upper normal level, Creatinine <1.25 x upper normal level. Albumin above lower normal level.
* Signed informed consent and expected cooperation of the patients for the treatment and followup must be obtained and documented according to GCP, and national/local regulations.
* All patients should have progressive disease according to RECIST-criteria, or intolerance to 1. line chemotherapy. Patients must be randomized before evaluation 8-12 weeks after starting 2. line chemotherapy.

Exclusion Criteria:

* Weight loss >10% the last 6 months
* Patient BMI > 30
* Previous resection of local relapse or non-hepatic metastasis within the last 2 years or resection of pulmonary or liver hilus lymph node metastases the last year.
* Previous diagnosed bone or CNS metastatic disease or thoracic or abdominal metastatic lymph nodes.
* Previous diagnosed cancer mammae or malignant melanoma.
* Non resected or palliative resection of primary CRC tumor.
* Liver metastases affecting the diaphragm determined by CT-scan and/or ultrasound examination.
* Liver lesion>10cm
* Three negative prognostic factors at time of randomization (CEA>80, less than 2 years from diagnosis, diameter of largest liver lesion >5.5cm).
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years from time of randomisation
  To determine overall survival after Ltx compared to palliative chemotherapy/other treatment in patients with progressive disease on chemotherapy or intolerance to 1-line chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Smedman, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway